CLINICAL TRIAL: NCT01971450
Title: Prospective Multicentre Non-interventional Study on Compliance of Inhaled Treatment With Ventavis in Patient With Pulmonary Hypertension
Brief Title: Non-interventional Study on Compliance of Inhaled Treatment With Ventavis in Patient With Pulmonary Hypertension
Acronym: IVENT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16777; VE1311RU (Other: Company internal)
Record Dates: First submitted 2013-09-20; First posted 2013-10-29 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Hypertension, Pulmonary
Keywords: Non-interventional; Ventavis; Iloprost; Pulmonary hypertension; Compliance; Russian Federation
MeSH Terms: conditions — Hypertension, Pulmonary; Patient Compliance | interventions — Iloprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Iloprost: The patients with pulmonary hypertension with inhaled treatment with Ventavis according to routine practice meeting the criteria of inclusion.
  Interventions: Drug: Iloprost (Ventavis, BAYQ6256)

INTERVENTIONS:
Drug: Iloprost (Ventavis, BAYQ6256)

SUMMARY:
Local, prospective, multicenter, non-comparative, non-interventional, observational study. It is planed to assess compliance of patients with PH (pulmonary hypertension) with the physician's recommendation in real practice.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years old
* Diagnosis of PH
* Planned or current treatment with Ventavis (not more than 6 month)

Exclusion Criteria:

* Contraindications for the use of Ventavis in accordance with the local product information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients ≥ 18 years old with PH, treated with Ventavis and for which the inclusion and exclusion criteria are fulfilled, are eligible for enrolment into the study.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Number of days without any drug administration at all | Up to 12 months
Number of fully inhaled doses in relation to the total number of inhalations per day | Up to 12 months
Number of missed doses per day as recommended | Up to 12 months
Number of actually inhaled doses per day vs. the recommended number of inhalations - either as recommended by the treating physician or as recommended by the label | Up to 12 months

SECONDARY OUTCOMES:
6 minute walking distance test (MWDT) value | Up to 12 months
Score on dyspnea Borg CR (category ratio) 10 scale | Up to 12 months
Patients' quality of life, assessed by validated questionnaire | Up to 12 months
Assessment of the structural changes in the lungs using X-ray examination of the lungs | Up to 12 months
Assessment of the structural changes in the lungs using spirography | Up to 12 months
Assessment of lung haemodynamics using the data of echocardiography | Up to 12 months
Assessment of lung haemodynamics using the data of catheterization | Up to 12 months
Reason for omission of inhalation as assessed by the physician | Up to 12 months
Concomitant medication for other indications than pulmonary hypertension | Up to 12 months
Number of participants with adverse events (AEs) | Up to 12 months
Severity of AEs | Up to 12 months
AE relation to treatment | Up to 12 months
AE treatment | Up to 12 months
AE outcomes | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Russia